CLINICAL TRIAL: NCT06660472
Title: Relationship Between Core Muscles Endurance and Saliba's Postural Classification System in Patients With Chronic Mechanical Low Back Pain
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Eltelbany, principal investigator, Cairo University
Other Study IDs: Sara-008490
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Core Muscles; Endurance; Saliba's Postural Classification System; Low Back Pain, Mechanical
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to investigate the relationship between core muscles endurance and Saliba Postural Classification System in patients with chronic mechanical low back pain.

DETAILED DESCRIPTION:
chronic mechanical low back pain (CMLBP) is a significant health issue affecting 85-90% of the general and athletic population, causing a significant socioeconomic burden. This study aims to address functional deficits in patients with CMLBP, reducing the burden and improving care delivery and work performance. Core muscle dysfunction, particularly multifidus and transversus abdominus muscles, is found in patients with CMLBP. However, the relationship between posture, function, and pain is not established due to the absence of a standardized postural classification system. The proposed tests can help infer the stability and function of core muscles in patients with CMLBP, enabling researchers to develop effective treatment programs. This study may also benefit physical therapists by providing an evidence-based approach in assessment using a valid and reliable postural classification system. Future research may address the relationship between core muscle endurance and Saliba Postural Classification System in patients with CMLBP.

ELIGIBILITY:
Inclusion Criteria:

1. Sixty male and female patients with CMLBP of more than 3 months duration
2. Patients with body mass between 18-25
3. Patients aged between 20-50 years old
4. Moderate level of pain (4-6 on visual analogue scale)
5. Minimal level of disability (0% to 20%) on Oswestry disability index as defined as "the patient can cope with most living activities. Usually, no treatment is indicated apart from advice on lifting, sitting, and exercise.

Exclusion Criteria:

Participants will be excluded if they did not meet the inclusion criteria mentioned above.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study was a cross sectional, Observational, and correlation analysis
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
assessment of pain intensity using visual analogue scale | at baseline
  The visual analog scale (VAS) is a unidimensional measure of pain intensity, consisting of a horizontal line 10 cm long. It is anchored by "no pain" (score 0) and "worst imaginable pain" (score 10), with higher scores indicating greater pain intensity.

SECONDARY OUTCOMES:
assessment of functional disability using cross-culturally adapted Arabic version of the Oswestry disability questionnaire | at baseline
  For each item of the ODI, the participants will be asked to choose one answer that best defines his/her back function. Scores for each item will be tallied and the total score will be recorded. A total score from 0-20 to indicate "minimal disability", 20-40 to indicate "moderate disability," 40-60 to indicate "severe disability", 60-80 to indicate "housebound", and 80-100 to indicate "bedbound".
assessment of mechanical stress points using vertical stress test to confirm the Saliba Postural Classification System | at baseline
  The patient is positioned on a stool, chair, or table, with their forearms vertically and hovering. Force is directed towards the patient, ensuring they cannot move unless they buckle. The therapist's hands are placed on the patient's shoulders between the acromion and the first rib insertion. The test is graded 1-5, with 1-4 indicating dysfunction and 5 being efficient force translation to the support base. Inefficient responses cause spine side bends, backward bends, shears, or rotates.
assessment of proper timing of core and global muscles in response to an external load using Elbow flexion test | at baseline
  The patient's position is described as a 90-degree bend in elbows, with forearms supinated to a loose pack position, humerus perpendicular to the floor, and no shoulder adduction allowed. The therapist's position involves standing in front, applying resistance, positioning forearms perpendicular to the floor, and hovering with hand placement over the distal end of the forearm. The patient's stability response is observed, with efficient states activating core, rotator cuff, shoulder girdle, and global shoulder and arm muscles. Inefficient states involve giving in arms, shoulder girdle, and spine.
assessment of trunk endurance using Trunk flexion test | at baseline
  The patient is positioned in a sit-up position with their back against a 60-degree jig, knees and hips flexed 90 degrees, arms folded, and feet secured. The therapist pulls the jig back 10 cm and the patient holds an isometric posture for as long as possible. Failure is determined when any part of the back touches the jig. The patient's time holding the isometric posture is recorded, with a normal range of 1-2 minutes.
assessment of back extensors (the erector spinae and the multifidus) endurance using trunk extension test | at baseline
  The back extensors, erector spinae and multifidus, are tested with the upper body off the bench and secured, with the pelvis, knees, and hips secured. Participants hold the upper limbs across the chest, and failure occurs when the upper body drops below the horizontal position. The researcher records the time participants can hold the body straight.
assessment of trunk side flexor endurance using side blank test | at baseline
  The test start with patient lying on the side then the therapist will ask him to lift the body on the elbow, forearm, and feet stacked creating a straight line from head to toe. Same as prone plank time recorded as long as he could hold his body and hip off the floor. The researcher will record the time with a normal range of 1-2 minute
assessment of trunk endurance using Prone plank test | at baseline
  The test start with the patient in prone position and the therapist will ask the patient to support the upper body off the ground by the elbows and forearms, and to take the weight by the toes with the legs straight. The hip is lifted off the floor creating a straight line from head to toe. As soon as the patient is in the correct position, the therapist starts the stopwatch. The head should be facing towards the ground and not looking forwards. The test is over when the patient is unable to hold the back straight and the hip is lowered. The researcher will record the time of holding the body up, normal range is 1-2 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Cairo university, Giza, Egypt